CLINICAL TRIAL: NCT04307017
Title: Physical Fitness Training Using Whole-Body Electrical Muscle Stimulation Among Individuals Living With Chronic Spinal Cord Injury
Brief Title: Fitness Training Using WBEMS Among Individuals With SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-5246
Record Dates: First submitted 2020-03-05; First posted 2020-03-13 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Spinal Cord Injuries
Keywords: Physical Fitness; Whole body electrical muscle stimulation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: StimaWell®EMS — The StimaWell®EMS device is a 12-channel medium-frequency device with modulated low frequency using a high-tech stimulation suit for the trunk and strap electrodes for the arms and legs allowing whole-body stimulation. The device has 70 preprogramed training programs based on goals (e.g., strengthening, endurance training, aerobic training).

SUMMARY:
Up to 15 individuals living with chronic SCI will be recruited for this study. Each participant will complete an initial clinical assessment before starting a 10-week training program. The training program will consist of three 45-minute Whole-Body Electrical Muscle Stimulation (WBEMS)-augmented exercise training sessions for 10 weeks. At each training session, all adverse events (pain, redness, injury, etc.) will be recorded along with participants' comments concerning comfort (i.e. Objective 1). The investigators hypothesize that the use of a WBEMS will result in no serious adverse effect during and following the training sessions and that it will take less than 10 minutes to don and doff the suit.

At the fifth session, after participants have had the opportunity to become familiar with the WBEMS intervention, the immediate effects of the intervention on physiological responses will be assessed (i.e. Objective 2). It is hypothesized that during a single training session consisting of WBEMS and exercise, physiological responses and energy expenditure (EE) will be significantly improved in participants with SCI compared to a training session consisting solely of exercises without WBEMS.

At the end of the training program, participants will complete the final clinical assessment to evaluate the therapeutic benefit of the WBEMS-augmented exercise intervention (i.e. Objective 3). Three months after the end of the training program, the participants will be asked to complete a semi-structured interview and questionnaire to evaluate the perceived benefits of the training program (i.e. Objective 3).It is also hypothesized that participants will perceive benefits of the 10-week training program such as decreased spasticity, increased energy and improved mood.

ELIGIBILITY:
Inclusion Criteria:

1. have a motor complete SCI (i.e., American Spinal Injury Association Impairment Scale grade A or B which means complete motor paralysis below the level of injury) at the neurological level T7 or below (i.e., to avoid triggering autonomic dysreflexia). The participants will have complete motor function of their arms but not of their legs;
2. be at least one year post-injury (i.e., chronic injury);
3. be between 18 and 65 years of age;
4. be cleared for physical activity based on The Physical Activity Readiness Questionnaire for Everyone (PAR-Q+)34
5. be able to provide informed, written consent.

Exclusion Criteria:

1) Contraindications for EMS35,36. Electrical stimulation should not be applied:

* if implanted electronic devices, including cardiac pacemakers
* if coronary stents are present
* if cosmetics and other implants are present in the application region
* to pregnant women
* on the regions of known or suspected malignancy
* if active deep vein thrombosis or thrombophlebitis
* to actively bleeding tissue or to persons with untreated hemorrhagic disorders
* to infected tissues, tuberculosis, or wounds with underlying osteomyelitis
* if inflammation is present in the region of application
* to recently radiated tissues
* to the chest in persons with cardiac disease, arrhythmias, or heart failure
* to the neck or head region of persons known to have seizures
* transcranially without specialized training
* to areas near reproductive organs or genitalia without specialized training
* to areas near or over eyes
* to anterior neck or carotid sinus
* to damaged or at-risk skin areas that would result in uneven conduction of current (excluding open wounds where the specific intent is to use electrical stimulation for tissue healing)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Duration of Training Session | For the 30 training sessions spread over 10 weeks
  Time in minutes
Intensity of Training Session | For the 30 training sessions spread over 10 weeks
  Type of activity; repetitions; weight resistance
Adverse Events | For the 30 training sessions spread over 10 weeks, if necessary
  All adverse events, even minor, will be reported in the intervention CRF, and compiled in a specific document (Adverse Event Report Form) all along the study to be analyzed as an outcome of the study

SECONDARY OUTCOMES:
Weight | Up to 10 weeks
Height | Up to 10 weeks
Body Mass Index | Up to 10 weeks
Anthropometric data | Up to 10 weeks
  Circumference of the waist, abdominal region, thighs, legs, arms and forearms
Maximal Isometric Voluntary Strength | Up to 10 weeks
  Maximal strength of the major muscle groups of upper extremity (i.e., flexors, extensors and abductors of the shoulder, and flexors and extensors of the elbow) will be measured using hand-held dynamometer
Exercise Self-Efficacy Questionnaire | Up to 10 weeks
  Used to assess the perception and confidence to do leisure time physical activity

CONTACTS AND LOCATIONS:
Locations (1):
- Lyndhurst Centre, Toronto Rehabilitation Institute-UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No